CLINICAL TRIAL: NCT00745485
Title: A Phase IV Study of the Safety and Feasibility of Rooms-based Infusion of Zoledronic Acid for Women With Post-menopausal Osteoporosis
Brief Title: Feasibility of Doctors' Rooms-based Infusion of Zoledronic Acid
Acronym: LISA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Clinical Disclosure Office, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446HAU27
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; zoledronic acid; postmenopausal women
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

ARMS (1):
- Zoldronic (Experimental)
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
1. The study will assess the safety and tolerability of a single-infusion of zoledronic acid 5 mg administered in a private medical practice setting by a nurse provided by a nationwide infusion service. Safety data will largely be monitored by investigating changes in the patients' well-being during the study.
2. The study will pilot and test a Patient Registry and Infusion Service process, which will allow zoledronic acid to be administered to trial patients in the investigators' private rooms by a team of roving nurses.

ELIGIBILITY:
Inclusion Criteria:

1. Female after menopause with osteoporosis either: 70 years of age or older with a bone mineral density T-score of -3.0 or less OR with a fracture due to minimal trauma.

Exclusion Criteria:

1. Intravenous bisphosphonate within the past 12 months
2. Abnormal levels of protein in the urine via dipstick at screening if not caused by bacterial infection
3. Abnormal liver function tests greater than twice normal
4. Evidence of high bone turnover
5. Abnormal calcium blood levels
6. Low Vitamin D levels
7. Poor renal function
8. Abnormal parathyroid function or uncontrolled, abnormal thyroid function
9. History of eye inflammation
10. History of diabetes leading to kidney or eye problems
11. A history of cancer except some non-invasive cancers of skin, colon, breast and cervix
12. Patients with severe dental problems or current dental infections Or requiring dental surgery
13. Known sensitivity to zoledronic acid or bisphosphonates

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 186 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | at baseline and month 12
Bone turnover | at baseline and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (14):
- Australia (14):
  - Novartis Investigative Site, Blacktown, New South Wales
  - Novartis Investigative Site, Georgetown, New South Wales
  - Novartis Investigative Site, Leichhardt, New South Wales
  - Novartis Investigative Site, Manly, New South Wales
  - Novartis Investigative Site, North Parramatta, New South Wales
  - Novartis Investigative Site, Wentworthville, New South Wales
  - Novartis Investigative Site, Caloundra, Queensland
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Ashford, South Australia
  - Novartis Investigative Site, Norwood, South Australia
  - Novartis Investigative Site, Footscray, Victoria
  - Novartis Investigative Site, Ringwood, Victoria
  - Novartis Investigative Site, Nedlands
  - Novartis Investigative Site, Nedlands Perth